CLINICAL TRIAL: NCT05764655
Title: Comparison of Troponin Assay With New POCT Method and in the Automation in the Decision-making Pathway of Patient With Chest Pain Suspected of Acute Myocardial Ischemia Entering the Emergency Room (POCT)
Brief Title: Comparison of Troponin Assay With New POCT Method in the Decision-making Pathway of Patient With Chest Pain Suspected of Acute Myocardial Ischemia in Emergency Room (POCT)
Acronym: POCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Sponsor
Other Study IDs: CCM 1720
Record Dates: First submitted 2023-02-21; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Chest Pain; Myocardial Ischemia
Keywords: chest pain; Myocardial Ischemia; POCT; Troponin
MeSH Terms: conditions — Chest Pain; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Troponin determination
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study aiming to evaluate the diagnostic accuracy of the high-sensitivity Troponin assay performed with the Atellica VTLi POCT system (by comparison with the results obtained with the Atellica diagnostic system currently in use) and to evaluate the impact of the POCT system on the reduction of decision-making time (particularly of "rule-out"), by evaluating the number of cases in which the conclusion of the decision pathway at 3 h (algorithm currently in use) could have been concluded at 1 h.

DETAILED DESCRIPTION:
Patients accessing the emergency room for chest pain suspected of acute myocardial ischemia, who are asked for Troponin determination for the decision pathway, will be asked to participate at the study. A blood draw will be performed (for determination of Troponin value, with classical method in use and with POCT method) at time:

* Zero (acess at the emergency room)
* 1 h
* 3 h

ELIGIBILITY:
Inclusion Criteria:

* Emergency department access for acute non-traumatic chest pain suspected of myocardial ischemia
* Sign of Informed Consent

Exclusion Criteria:

* Diagnostic electrocardiographic picture for Acute Coronary Syndrome-STEMI (ACS-STEMI)
* Absence of symptomatology in the 12 hours prior to admission to the emergency room
* Post-traumatic chest pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients accessing at emergency room for acute chest pain suspected of acute myocardial ischemia, who are asked for Troponin determination in the pathway decision-making.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of the high-sensitivity Troponin assay performed with the Atellica VTLi POCT system | through study completion, an average of 1 year
  Evaluate the diagnostic accuracy of the high-sensitivity Troponin assay performed with the Atellica VTLi POCT system by comparison with results obtained with the Atellica diagnostic system currently in use

SECONDARY OUTCOMES:
The impact of the POCT system on the reduction of decision-making time | through study completion, an average of 1 year
  Evaluate the impact of the POCT system on the reduction of decision-making time, by evaluating the number of cases in which the end of the decision pathway at 3 h (algorithm currently in use) could have been done at 1 h

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Biondi, MD, PhD, Principal Investigator — IRCCS Centro Cardiologico Monzino
Locations (1):
- IRCCS Centro Cardiologico Monzino, Milan, Italy